CLINICAL TRIAL: NCT07099456
Title: Channelling Fertility And Sexual Function In Congenital Adrenal Hyperplasia. CALLIOPE: An Observational, Longitudinal Pilot Study
Brief Title: Fertility And Sexual Function In CAH: CALLIOPE
Acronym: CALLIOPE
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Federico II University (Other); S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor of Endocrinology and Metabolism, University of Roma La Sapienza
Other Study IDs: CALLIOPE
Record Dates: First submitted 2025-07-02; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Congenital Adrenal Hyperplasia (CAH)
Keywords: congenital adrenal hyperplasia; CAH; fertility; LC-MS/MS; semen analysis; reproductive function
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, saliva, urine and semen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Congenital Adrenal Hyperplasia (CAH): Adult patients with a known/new diagnosis of CAH requiring chronic glucocorticoid replacement therapy

SUMMARY:
This is a multicenter study designed to assess the effects of groundbreaking CAH therapies on a spectrum of clinical and biochemical outcomes, with a special emphasis on reproductive and sexual health. Fertility is a profound concern for individuals with CAH, given the high prevalence of gonadal dysfunction that arises from the hormonal derangements that characterize this complex disease. At our endo-ERN accredited center for rare diseases at Policlinico Umberto I, addressing these fertility issues in CAH patients represents a daily commitment. The revolution of the pharmacological management of CAH is one of the most debated topics to date. Data on the effects of novel management options for CAH on fertility are scarce, but the anecdotal improvements in sperm count and menstrual regularity reported in the latest clinical trials have significantly motivated us to design the CALLIOPE study. Thus, we aim to delve deeper into the fertility and sexual function of CAH patients, employing advanced seminal parameter evaluations, multiparametric gonadal ultrasound, and sophisticated hormonal analyses in both females and males performed by ultra-high performance liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS). Beyond fertility, the CALLIOPE trial aspires to provide further understanding of therapy's effects on body composition, metabolism, immune function, coagulation, and quality of life, among other factors. We will explore the immunological impact of novel CAH therapies by quantifying Peripheral Blood Mononuclear Cells (PBMCs) and analyzing transcriptomic profiles to unveil gene expression patterns and identify biomarkers that could signal therapeutic targets or disease management strategies in CAH. Moreover, seminal plasma will be used to assess the expression of adrenal miRNAs regulating steroidogenesis and metabolism.

The research will be conducted at our rare disease referral center (Policlinico Umberto I, Sapienza University of Rome) in collaboration with leading centers across Italy: Modena (Università degli Studi di Modena e Reggio Emilia), Naples (Università Federico II), Rome (Ospedale Sant'Andrea) and Bologna (Alma Mater Studiorum - Università di Bologna).

https://isidorilab.com/home

DETAILED DESCRIPTION:
Classic Congenital Adrenal Hyperplasia (CAH) is the most common rare disease affecting the adrenal glands. It is characterized by primary adrenal insufficiency due to congenital enzymatic defects, which impair glucocorticoid synthesis. As a result, patients require lifelong glucocorticoid replacement therapy, often combined with mineralocorticoid supplementation in the salt-wasting form of the disease. Standard treatment involves short-acting, immediate-release glucocorticoids (such as hydrocortisone or cortisone acetate) administered two or three times daily. Although lifesaving, chronic glucocorticoid therapy is associated with increased cardiometabolic risk, altered glucose and lipid metabolism, weight gain, osteoporosis, higher infection susceptibility, and reduced life expectancy, even at replacement-level doses.

In CAH, supraphysiologic doses and reverse circadian timing of glucocorticoid administration are often employed to suppress androgen excess. This approach, however, may exacerbate side effects related to glucocorticoid overexposure. A dose-dependent impact of glucocorticoid therapy has been observed on cardiovascular risk, bone mineral density, body composition, and immune function. Despite these known effects, reproductive and sexual health outcomes remain under-investigated, representing a significant unmet need in the comprehensive management of CAH.

In male patients, reproductive dysfunction is frequently observed and is often attributed to the development of testicular adrenal rest tumors (TARTs), which can impair fertility. Current medical approaches to TARTs include high-dose, long-acting glucocorticoid therapy, with variable effects on tumor regression and semen quality. However, this strategy is associated with additional metabolic and cardiovascular risks. Furthermore, uncontrolled androgen excess may be converted to estrogens and, together with elevated progestogen levels, suppress the hypothalamic-pituitary-gonadal axis, contributing to hypogonadotropic hypogonadism.

Female patients with CAH may present with menstrual disturbances, anovulation, biochemical and clinical hyperandrogenism, and infertility. Additionally, non-hormonal factors such as anatomical variations and psychological distress may impact sexual health and reproductive intentions.

Recent advances in CAH therapy include the development of novel glucocorticoid formulations that aim to better replicate the circadian rhythm of cortisol secretion. Dual-release hydrocortisone and non-glucocorticoid therapeutic options have shown promise in improving metabolic, immunological, and hormonal parameters, and may allow a decoupling of glucocorticoid replacement from androgen suppression. However, real-world data on the long-term cardiometabolic outcomes of these newer treatments remain limited, and reproductive parameters-such as semen quality, pregnancy rates, and menstrual cycle normalization-require further clinical investigation.

The aim of this observational prospective study is to evaluate the impact of hormonal alterations and treatment strategies on reproductive and sexual health in individuals with CAH. The study will adopt a multidimensional clinical-translational approach, integrating clinical assessments with advanced profiling techniques such as steroidomics, microRNA analysis, and gene expression profiling. These precision medicine tools are expected to identify novel biomarkers and mechanistic pathways involved in reproductive dysfunction, ultimately supporting the development of targeted therapeutic strategies.

Following screening based on inclusion and exclusion criteria, eligible participants will provide informed consent and undergo baseline evaluations. Follow-up assessments will be conducted after significant modifications in therapy or lifestyle interventions, typically within 3 to 6 months. In the absence of changes, at least one follow-up evaluation will be scheduled within a 3- to 12-month timeframe, as appropriate for each participant. Study evaluations will be integrated into routine clinical care without altering standard management protocols.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, males in the age range 18-65 years and pre-menopausal females in the age range 18-55 years;
* a known/new diagnosis of CAH.

Exclusion Criteria:

* BMI > 40 Kg/m2;
* Any other concomitant condition requiring steroid treatment;
* Severe liver and/or kidney disease;
* Thyroid dysfunctions (overt hyperthyroidism and hypothyroidism);
* Malignant neoplasms;
* Drug and alcohol abuse;
* Use of drugs acting on hormonal levels (e.g. antiandrogens);
* Psychiatric diseases;
* Postmenopausal women;
* Women taking combined oral contraceptive pill (women) or other contraceptives will require stability for at least 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with congenital adrenal hyperplasia (CAH) under glucocorticoid treatment
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in sperm concentration (total count per ejaculate) at semen analysis (male subjects) | At baseline and during follow-up (up to 5 years)
  Sperm concentration will be evaluated through standard semen analysis in male participants, according to WHO guidelines.
  Measurements will be used to assess changes over time in relation to disease control and treatment modifications. Semen analyses will be repeated at follow-up visits if clinically indicated or in case of significant therapeutic changes.
  Unit of Measure: millions per ejaculate (10⁶/ejaculate)
Change in sperm concentration (concentration per mL) at semen analysis (male subjects) | At baseline and during follow-up (up to 5 years)
  Sperm concentration will be evaluated through standard semen analysis in male participants, according to WHO guidelines.
  Measurements will be used to assess changes over time in relation to disease control and treatment modifications. Semen analyses will be repeated at follow-up visits if clinically indicated or in case of significant therapeutic changes.
  Unit of Measure: millions per mL (10⁶/mL)
Change in Serum Testosterone:LH ratio (female subjects) | At baseline and during follow-up (up to 5 years)
  Assessment of changes in the ratio between serum total testosterone and luteinizing hormone (LH) concentrations in female participants. Blood samples will be collected in the early follicular phase or as appropriate based on menstrual status. The ratio will be calculated at each time point, and changes will be expressed as percent change from baseline or through paired comparison.
  The aim is to evaluate this ratio as a potential biomarker of hyperandrogenism severity and treatment response.
  Unit of Measure: Ratio (ng/dL per IU/L)
Change in serum Estradiol:FSH ratio (female subjects) | At baseline and during follow-up (up to 5 years)
  Evaluation of changes in the ratio between serum estradiol (E2) and follicle-stimulating hormone (FSH) concentrations in female participants. Blood samples will be collected in the early follicular phase when possible or based on clinical context. The E2:FSH ratio will be calculated at each visit and used to assess hypothalamic-pituitary-ovarian axis function and treatment effects over time. Changes will be analyzed using paired comparisons or percentage variation from baseline.
  This outcome is part of a broader hormonal assessment that includes additional ratios such as Testosterone:LH.
  Unit of Measure: Ratio (pg/mL per mIU/mL)

SECONDARY OUTCOMES:
Number of pregnancies and childbirths from baseline | From baseline until the end of the study (up to 5 years)
  For female participants and for partners of male participants who express the intention to conceive, data on the occurrence of pregnancies and childbirths will be collected during the study period. Outcomes will be reported as absolute numbers of confirmed pregnancies and live births. This measure aims to assess reproductive outcomes in patients with CAH under different treatment regimens.
  Unit of Measure: Count (number of pregnancies and number of childbirths)
Change in bilateral testicular volume and TARTs volume (scrotal ultrasound, male subjects) | At baseline and during follow-up (up to 5 years)
  Evaluation of bilateral testicular volume and testicular adrenal rest tumor (TART) volume in male participants, assessed via standardized scrotal ultrasound. Volumes will be calculated using the ellipsoid formula:
  Volume = width × depth × length × 0.52
  Measurements will be recorded at each visit to monitor anatomical changes over time and assess the response to clinical management. Unit of Measure: volume (mL)
Change in fructose levels in seminal plasma (male subjects) | At baseline and during follow-up (up to 5 years)
  Biochemical evaluation of seminal plasma in male participants, specifically measuring fructose concentration. This marker reflects the function of seminal vesicles and prostate, and may provide indirect information on androgen status and reproductive function.
  Unit of Measure: mg/dL
Change in Circadian, multi-matrix, serum, urinary and salivary LC-MS/MS steroid profiles | At baseline and during follow-up (up to 5 years)
  * From blood samples taken at 8 AM, 12 AM, 4 PM and 8 PM, several steroids including glucocorticoids, mineralocorticoids, androgens, and their precursors and metabolites will be evaluated;
  * 24-hours urine samples will be used to evaluate several steroids and their metabolites and to estimate enzyme activities (11β-Hydroxysteroid dehydrogenase type 1/2, 5α-reductase)
  * All patients will collect at their home saliva samples at 8 AM, 10 AM, 12 PM, 4 PM, 6 PM, 8 PM and 12 AM. Saliva samples will be used to assess steroid metabolism.
  Unit of measure: ng/mL for all steroids
Change in Circadian quantification of Peripheral Blood Mononuclear Cells (PBMCs) subpopulations by flow cytometry | At baseline and during follow-up (up to 5 years)
  From blood samples taken at 8 AM, 12 AM, 4 PM and 8 PM, a quantification of the distribution of peripheral blood mononuclear cell (PBMC) subpopulations will be performed using multicolor flow cytometry. Cell populations assessed will include, but are not limited to, T cells, B cells, NK cells, and monocytes. The goal is to evaluate circadian variation and treatment-related changes in immune cell composition.
  Unit of measure: Percentage of total PBMCs (%)
Change in total and regional fat and lean mass measured by DXA | At baseline and during follow-up (up to 5 years)
  Dual X-ray Absorptiometry (DXA) will be used to assess total and segmental fat mass and lean mass (trunk, arms, legs). This outcome will monitor changes in body composition over time in relation to disease status and therapeutic interventions. Unit of measure: Mass (grams or kilograms)
Change in Bone mineral density (BMD) of femur and lumbar spine assessed by DXA | Baseline and follow-up scans every 18-24 months, until the end of the study (up to 5 years)
  Bone mineral density (BMD) will be measured at the femoral neck and lumbar spine using Dual X-ray Absorptiometry (DXA). Values will be used to monitor bone health and assess changes over time in relation to glucocorticoid therapy and disease management.
  Unit of Measure: Grams per square centimeter (g/cm²)
Change in International Index of Erectile Function (IIEF-15) questionnaire score (male sexual dysfunction) | At baseline and during follow-up (up to 5 years)
  The International Index of Erectile Function (IIEF-15) questionnaire will be administered to male participants to assess erectile function and broader aspects of sexual health. The total score and individual domain scores (erectile function, orgasmic function, sexual desire, intercourse satisfaction, overall satisfaction) will be evaluated at each time point to monitor sexual dysfunction and its changes over time.
  Unit of Measure:
  IIEF-15 score (range: 5-75)
Change in Structural cardiac parameters assessed by transthoracic echocardiography | At baseline and during follow-up (up to 5 years)
  Cardiac structural dimensions will be measured by transthoracic echocardiography and will include:
  Left ventricular end-diastolic diameter (LVEDD)
  Left ventricular end-systolic diameter (LVESD)
  Interventricular septum thickness (IVS)
  Posterior wall thickness (PW)
  Epicardial fat thickness (EFT)
  These measurements will assess cardiac remodeling and visceral fat accumulation.
  Unit of Measure: Millimeters (mm)
Change in Lipid metabolism parameters | At baseline and during follow-up (up to 5 years)
  Evaluation of lipid profile and associated biomarkers, including:
  Total cholesterol;
  High-density lipoprotein cholesterol (HDL-c);
  Triglycerides;
  Calculated low-density lipoprotein cholesterol (LDL-c);
  Non-HDL cholesterol;
  Apolipoproteins A and B.
  These values will be measured from fasting blood samples and used to assess cardiovascular risk and metabolic health.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in CAHQoL questionnaire scores (Health-related Quality fo Life) | At baseline and during follow-up (up to 5 years)
  Health-related quality of life (HRQoL) specific to congenital adrenal hyperplasia (CAH) will be evaluated using the CAH-QoL questionnaire, a disease-specific validated tool. The total score and subdomain scores will be recorded and analyzed over time.
  Unit of Measure: CAH-QoL total score (range: questionnaire-specific, higher scores indicate better HRQoL)
Change in Serum liver enzymes (AST, ALT, gamma-GT, alkaline phosphatase) | At baseline and during follow-up (up to 5 years)
  Description: Measurement of serum levels of AST (GOT); ALT (GPT); gamma-glutamyl transferase (gamma-GT); and alkaline phosphatase to evaluate liver function.
  Unit of Measure: Units per liter (U/L)
Change in total sperm motility (& motile spermatozoa) at semen analysis (male subjects) | At baseline and during follow-up (up to 5 years)
  Description: - Changes (%change and paired analysis) in the percentage of total motile spermatozoa
Change in the percentage of spermatozoa with typical morphology at semen analysis (male subjects) | At baseline and during follow-up (up to 5 years)
  Changes in the percentage of spermatozoa with typical morphology at semen analysis
Change from Baseline in Number of Regular Menses (female subjects) | during follow-up (up to 5 years)
  Evaluation of the change in menstrual frequency, defined as the number of spontaneous, regular menses occurring per calendar month. Regular menses are defined as occurring every 21-35 days. Information on the menses will be collected by the patients in a menstrual diary.The outcome will assess restoration or maintenance of normal menstrual patterns over time.
Change in Testicles and TARTs vascularity (Testicular Ultrasound, male subjects) | At baseline and during follow-up (up to 5 years)
  Vascularity will be assessed at testicular ultrasound and will be scored based on the operator evaluation as follows:
  0: absent vascularity
  1. normal vascularity
  2. increased vascularity
  3. very increased vascularity
Change in Testicles and TARTs parenchymal homogeneity (Testicular Ultrasound, male subjects) | At baseline and during follow-up (up to 5 years)
  Homogeneity will be assessed at testicular ultrasound and will be scored based on the operator evaluation as follows:
  0: homogeneous echo-texture
  1. mild inhomogeneous echo-texture
  2. inhomogeneous echo-texture
  3. severe inhomogeneous echo-texture
Change in TARTs number (Testicular Ultrasound, male subjects) | At baseline and during follow-up (up to 5 years)
  TARTs number will be evaluated as count (n)
Change in Radiomic features of testicular adrenal rest tumors (TARTs) and normal testicular parenchyma on ultrasound imaging | At baseline and during follow-up (up to 5 years)
  Quantitative extraction and comparison of radiomic features from grayscale and Doppler ultrasound images of TARTs and contralateral normal testicular parenchyma. Features will include first-order statistics (e.g., intensity histograms), texture metrics (e.g., GLCM, GLRLM), and shape descriptors. The analysis aims to identify imaging biomarkers associated with lesion vascularization, composition, and potential progression.
  Radiomic features will be extracted using standardized algorithms and open-source platforms (e.g., PyRadiomics). Images will be manually segmented by trained observers, with interobserver variability assessed. The goal is to assess whether radiomics can differentiate TARTs from healthy tissue and monitor response to therapy over time.
  Unit of measure: Dimensionless radiomic feature values (e.g., entropy, kurtosis, contrast, etc.)
Change in CEUS perfusion patterns (time parameters) of testicular adrenal rest tumors (TARTs, male participants) and other testicular inhomogeneities | At baseline and during follow-up (up to 5 years)
  Assessment of perfusion characteristics of TARTs and testicular inhomogeneities using contrast-enhanced ultrasound (CEUS). Quantitative CEUS parameters (e.g., time to peak, wash-in and wash-out times) will be extracted and analyzed at baseline and during follow-up. The aim is to evaluate changes in tumor vascularity in response to treatment or disease evolution.
  Unit of Measure: Time (seconds)
Change in Anthropometric Parameters | At baseline and during follow-up (up to 5 years)
  Assessment of anthropometric parameters including:
  Height;
  Waist circumference;
  Hip circumference;
  Measurements will be performed using standardized protocols to evaluate body proportions and fat distribution.
  Unit of Measure: Centimeters (cm)
Change in CEUS perfusion patterns (intensityparameters) of testicular adrenal rest tumors (TARTs, male participants) and other testicular inhomogeneities | At baseline and during follow-up (up to 5 years)
  Assessment of perfusion characteristics of TARTs and testicular inhomogeneities using contrast-enhanced ultrasound (CEUS). Quantitative CEUS parameters (peak intensity) will be extracted and analyzed at baseline and during follow-up. The aim is to evaluate changes in tumor vascularity in response to treatment or disease evolution.
  Unit of Measure: signal intensity (arbitrary units, AU) per CEUS software analysis
Change in ovarian volume (pelvic ultrasound, female subjects) | Baseline and follow-up visits (up to 5 years)
  Description
  Evaluation of ovarian volume in female participants using pelvic ultrasound. Measurements will be taken for both ovaries using the ellipsoid formula:
  Volume= width × depth × length × 0.52 Data will be used to assess changes over time in relation to hormonal status and treatment response.
  Unit of Measure: Cubic centimeters (cm³)
Change in number of ovarian follicular cysts (pelvic ultrasound, female subjects) | At baseline and during follow-up (up to 5 years)
  Pelvic ultrasound will be used to evaluate the number of follicular cysts in each ovary. This outcome will monitor changes potentially associated with androgen excess and ovulatory function.
  Unit of Measure: Number of cysts (count)
Change in size of ovarian follicular cysts (pelvic ultrasound, female subjects) | At baseline and during follow-up (up to 5 years)
  Pelvic ultrasound will be used to evaluate the diameter of follicular cysts in each ovary. This outcome will monitor changes potentially associated with androgen excess and ovulatory function.
  Unit of Measure: Maximum cyst size in millimeters (mm)
Change in Ultrasonographic signs of ovulation (pelvic ultrasound, female subjects) | At baseline and during follow-up (up to 5 years)
  Pelvic ultrasound will be used to assess indirect signs of ovulation, including corpus luteum appearance, follicular rupture, and mid-luteal phase changes. This outcome aims to monitor ovulatory status in relation to treatment and hormonal balance. Unit of Measure: Binary (ovulation detected: yes/no)
Presence of ovarian adrenal rest tumors (OARTs) on pelvic ultrasound | At baseline and during follow-up (up to 5 years)
  Evaluation of the presence or absence of ovarian adrenal rest tumors (OARTs) in female participants through pelvic ultrasound. If visualized, lesion characteristics such as size and echogenicity will also be recorded for exploratory purposes.
  Unit of Measure: Binary (present/absent)
Change in seminal acid phosphatase levels (male subjects) | At baseline and during follow-up (up to 5 years)
  Biochemical evaluation of seminal plasma in male participants, specifically measuring acid phosphatase activity. This marker reflects the function of seminal vesicles and prostate, and may provide indirect information on androgen status and reproductive function.
  Unit of Measure: Acid phosphatase: IU/L
Change in Expression levels of microRNAs in serum and seminal plasma (male subjects) | At baseline and during follow-up (up to 5 years)
  Next-generation sequencing (NGS) will be used to quantify the expression levels of circulating microRNAs (miRNAs) in both serum and seminal plasma of male participants. Global miRNA profiling will be performed, with downstream analyses including targeted evaluation of selected miRNAs of interest, such as miR-125a-5p, miR-320a-3p, let-7b, miR-132, and miR-455. Analyses aim to identify disease- or treatment-associated changes in miRNA expression over time.
  Unit of measure: Relative expression (normalized counts or fold change)
Change in Circadian transcriptomic profile of PBMCs using targeted gene expression analysis | At baseline and during follow-up (up to 5 years)
  Gene expression profiles of PBMCs will be assessed from samples collected at four circadian time points using NanoString technology. A predefined panel of 400 genes will be analyzed to evaluate circadian transcriptional patterns and their modulation by treatment. Expression data will be normalized and analyzed for circadian rhythm dynamics and pathway enrichment.
  Unit of measure: Normalized gene expression (counts or fold change)
Prevalence and incidence of asymptomatic vertebral fractures (lateral spine imaging, DXA) | Baseline and follow-up assessments every 18-24 months, until the end of the study (up to 5 years)
  Asymptomatic vertebral fractures will be evaluated through vertebral fracture assessment (VFA) or lateral spine imaging performed during DXA scans. Fractures will be classified according to semiquantitative or Genant criteria. The aim is to detect subclinical vertebral damage associated with chronic glucocorticoid exposure.
  Unit of Measure: Count (number of fractures)
Change in Trabecular Bone Score (TBS) calculated from lumbar spine DXA | Baseline and follow-up assessments every 18-24 months, until the end of the study (up to 5 years)
  Trabecular Bone Score (TBS) will be derived from lumbar spine DXA scans to assess bone microarchitecture. TBS is a dimensionless value reflecting trabecular texture, and will be used as an additional parameter to evaluate bone quality independently of BMD. Unit of measure: TBS index (dimensionless value)
Change in body composition indices and fat distribution ratios measured by DXA | At baseline and during follow-up (up to 5 years)
  From DXA scans, the following indices will be calculated:
  Total and appendicular lean mass index (lean mass/height²)
  Total and appendicular fat mass index (fat mass/height²)
  Android-to-gynoid fat mass ratio
  Trunk-to-limb fat mass ratio
  These parameters will be used to evaluate changes in body composition patterns and fat distribution associated with hormonal status and treatment. Unit of measure: Dimensionless ratios or indexed values (e.g., kg/m²)
Change in Left ventricular mass index (LVMI) assessed by echocardiography | At baseline and during follow-up (up to 5 years)
  LVMI will be calculated from transthoracic echocardiography measurements, indexed to body surface area, as a marker of left ventricular hypertrophy.
  Unit of Measure:
  Grams per square meter (g/m²)
Change in Left atrial volume index (LAVI) assessed by echocardiography | At baseline and during follow-up (up to 5 years)
  Left atrial volume index will be calculated and expressed as volume per body surface area, to assess atrial remodeling and diastolic function.
Change in Left ventricular ejection fraction (EF) assessed by echocardiography | At baseline and during follow-up (up to 5 years)
  Ejection fraction will be calculated to evaluate global systolic function of the left ventricle using Simpson's biplane method. Unit of Measure: Percentage (%)
Change in Doppler-derived diastolic function parameters (E/A and E/e' ratios) | At baseline and during follow-up (up to 5 years)
  Mitral inflow and tissue Doppler imaging will be used to calculate:
  E/A ratio (early-to-late ventricular filling velocity)
  E/e' ratio (early mitral inflow velocity to early mitral annular velocity)
  These values are markers of diastolic function and left ventricular filling pressures.
  Unit of Measure: Unitless ratios
Change in Fasting glucose and C-peptide levels (mg/dL) | At baseline and during follow-up (up to 5 years)
  Measurement of fasting glucose and C-peptide from venous blood samples to assess glycemic control and beta-cell activity.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in Fasting insulin levels (µU/mL) | At baseline and during follow-up (up to 5 years)
  Evaluation of fasting serum insulin levels to estimate insulin sensitivity and support HOMA-IR calculation.
  Unit of Measure: Micro-units per milliliter (µU/mL)
Change in Glycated hemoglobin (HbA1c) | At baseline and during follow-up (up to 5 years)
  Measurement of HbA1c to assess long-term glycemic control.
  Unit of Measure: Percentage (%)
Change in Insulin resistance index (HOMA-IR) | At baseline and during follow-up (up to 5 years)
  Description:
  Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) will be calculated from fasting insulin and glucose values to estimate peripheral insulin sensitivity.
  Unit of Measure: Dimensionless index
Change in Prothrombin time and activated partial thromboplastin time (seconds) | At baseline and during follow-up (up to 5 years)
  Assessment of blood clotting times using:
  Prothrombin time (PT);
  Activated partial thromboplastin time (aPTT);
  Used to evaluate the function of extrinsic and intrinsic coagulation pathways.
  Unit of Measure: Seconds
Change in International Normalized Ratio (INR) | At baseline and during follow-up (up to 5 years)
  Calculation of the INR value from prothrombin time to standardize coagulation monitoring across labs.
  Unit of Measure: INR (dimensionless ratio)
Change in Fibrinogen levels and coagulation factors (mg/dL) | At baseline and during follow-up (up to 5 years)
  Quantification of:
  Fibrinogen;
  Coagulation factors V, VII, VIII;
  Protein C;
  Protein S;
  Antithrombin.
  Measured from plasma to evaluate thrombotic risk and clotting factor levels.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in Coagulation factor activity (functional %) | At baseline and during follow-up (up to 5 years)
  Measurement of coagulation factor and anticoagulant protein activity expressed as a percentage of normal control, including:
  Factor V, VII, VIII activity;
  Protein C and S activity;
  Antithrombin activity.
  Unit of Measure: Percentage (%)
Change in FSFI-19 questionnaire score (female sexual dysfunction) | At baseline and during follow-up (up to 5 years)
  The FSFI-19 (Female Sexual Function Index - 19 items) will be used to assess sexual function in female participants. This self-administered, validated questionnaire evaluates six domains of female sexual function over the previous 4 weeks: Desire (items 1-2, score range 1.2-6.0); Arousal (items 3-6, score range 0-6.0); Lubrication (items 7-10, score range 0-6.0); Orgasm (items 11-13, score range 0-6.0); Satisfaction (items 14-16, score range 0.8-6.0); Pain (items 17-19, score range 0-6.0) Each domain score is obtained by multiplying the sum of the domain's item scores by a domain-specific factor. The total FSFI score is the sum of the six domain scores and ranges from 2.0 to 36.0. Higher scores indicate better sexual function. A score below the established cutoff (commonly 26.55) suggests risk of sexual dysfunction. This outcome will be used to track changes in sexual health status over time and in response to therapeutic interventions.
  Unit of Measure:FSFI-19 total score, range: 2-36
Change in body weight | At baseline and during follow-up (up to 5 years)
  Description:
  Assessment of body weight using calibrated scales under standardized conditions.
  Unit of Measure: Kilograms (kg)
Change in Body Mass Index | At baseline and during follow-up (up to 5 years)
  Calculation of body mass index (BMI = weight/height²), to assess general adiposity.
  Unit of Measure: Ratio (kg/m²)
Change in waist-to-hip ratio and waist-to-height ratio | At baseline and during follow-up (up to 5 years)
  Calculation of anthropometric ratios: waist-to-hip ratio (WHR = waist circumference/hip circumference) and waist-to-height ratio (WHtR ) waist circumference/height). These indicators are used to assess general and central adiposity.
  Unit of Measure: Dimensionless ratios
Change in blood pressure | At baseline and during follow-up (up to 5 years)
  Measurement of systolic and diastolic blood pressure in a seated and rested condition, using standard oscillometric or auscultatory methods.
  Unit of Measure: Millimeters of mercury (mmHg)
Change in Handgrip strength test | At baseline and during follow-up (up to 5 years)
  Description:
  Evaluation of muscle strength using a handgrip dynamometer. The best result of three trials with the dominant hand will be recorded.
  Unit of Measure: Kilograms (kg)
Change in Ferriman-Gallwey score (female subjects) | At baseline and during follow-up (up to 5 years)
  Description:
  Assessment of hirsutism in female participants using the Ferriman-Gallwey scoring system, based on hair distribution in nine androgen-sensitive body areas.
  Unit of Measure: Clinical score (0-36)
Change in Chair stand test (5-times sit-to-stand) and Balance test | At baseline and during follow-up (up to 5 years)
  Description:
  The 5-times sit-to-stand test will be used to assess lower limb strength and functional mobility. Participants will be asked to rise from a chair and sit down 5 times consecutively as quickly as possible without using their arms. Time to completion will be recorded using a stopwatch. Static balance will be assessed using standard balance tests, such as tandem, semi-tandem, or one-leg stand positions. Time maintained in each position without support will be recorded, and postural stability will be monitored.
  Unit of Measure: Seconds (s)
Change in Gait speed test | At baseline and during follow-up (up to 5 years)
  Gait speed will be assessed over a standardized distance (e.g., 4 or 6 meters), measuring the time taken to walk at a usual pace. Gait speed will be calculated to evaluate mobility, frailty, and risk of functional decline.
  Unit of Measure: Meters per second (m/s)
Change in Short Physical Performance Battery (SPPB) total score | At baseline and during follow-up (up to 5 years)
  The Short Physical Performance Battery (SPPB) will be used to assess lower extremity function in participants. The SPPB includes three components:
  Gait speed test over a short distance (e.g., 4 meters);
  Chair stand test (5-times sit-to-stand);
  Balance test (side-by-side, semi-tandem, and tandem stance).
  Each component is scored from 0 to 4, with a maximum total score of 12. Higher scores indicate better physical performance. The total SPPB score will be used to monitor functional status and identify early signs of physical frailty.
  Unit of Measure SPPB score (range: 0-12)
Change in AddiQoL questionnaire score (Health-related quality of life) | At baseline and during follow-up (up to 5 years)
  Description:
  Quality of life in the context of adrenal insufficiency will be evaluated using the AddiQoL questionnaire. This validated tool measures patient-reported well-being in those undergoing glucocorticoid replacement therapy. Total and domain-specific scores will be analyzed.
  Unit of Measure: AddiQoL score (range: questionnaire-specific, higher scores indicate better quality of life)
Change in Short Form 36 questionnaire score (General health-related quality of life) | At baseline and during follow-up (up to 5 years)
  Description:
  The Short Form 36 (SF-36) questionnaire will be used to assess general health-related quality of life across 8 domains: physical functioning; role limitations due to physical health; bodily pain; general health; vitality; social functioning; role limitations due to emotional problems; and mental health. A physical component score (PCS) and mental component score (MCS) will also be derived.
  Unit of Measure: SF-36 score (range: 0-100 per domain, higher scores indicate better quality of life)
Change in Pittsburgh Sleep Quality Index scores (PSQI) (Sleep quality) | At baseline and during follow-up (up to 5 years)
  Description:
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a validated questionnaire that assesses sleep disturbances over the previous month. It includes 7 components: subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleep medication; and daytime dysfunction. A global score will be calculated.
  Unit of Measure: PSQI total score (range: 0-21, higher scores indicate worse sleep quality)
Change in Serum bilirubin levels | At baseline and during follow-up (up to 5 years)
  Description: Total, direct, and indirect serum bilirubin concentrations will be measured to assess liver excretory function.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in Serum creatinine | At baseline and during follow-up (up to 5 years)
  Description: Evaluation of kidney function through measurement of serum creatinine.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in Urinary creatinine and electrolytes (24-hour collection) | At baseline and during follow-up (up to 5 years)
  Description: Measurement of creatinine and electrolytes (sodium, potassium, chloride, calcium) in 24-hour urine samples to evaluate renal excretion.
  Unit of Measure: Milligrams per 24 hours (mg/24h) or millimoles per liter (mmol/L)
Change in Serum levels of Inhibin B and SHBG | At baseline and during follow-up (up to 5 years)
  Description: Measurement of reproductive hormone markers: inhibin B and sex hormone-binding globulin (SHBG).
  Unit of Measure: Nanograms per milliliter (ng/mL)
Change in Serum C Reactive Protein | At baseline and during follow-up (up to 5 years)
  Description: Measurement of systemic inflammation through C-reactive protein (CRP) Unit of Measure: Milligrams per liter (mg/L)
Change in erythrocyte sedimentation rate (ESR) | At baseline and during follow-up (up to 5 years)
  Description: Measurement of systemic inflammation through erythrocyte sedimentation rate (ESR).
  Unit of millimeters per hour (mm/h) for ESR
Change in Serum albumin | At baseline and during follow-up (up to 5 years)
  Measurement of serum albumin concentration as a marker of nutritional and protein status.
  Unit of Measure: Grams per deciliter (g/dL)
Change in Plasma levels of POMC-derived peptides | At baseline and during follow-up (up to 5 years)
  Description: Measurement of POMC-related peptides in plasma samples (e.g., ACTH, α-MSH), analyzed by immunoassays.
  Unit of Measure: Picograms per milliliter (pg/mL)
Change in Serum TSH levels | At baseline and during follow-up (up to 5 years)
  Measurement of thyroid-stimulating hormone (TSH) in serum to evaluate pituitary-thyroid axis activity.
  Unit of Measure: International units per liter (IU/L)
Change in Serum free T3 (fT3) levels | At baseline and during follow-up (up to 5 years)
  Measurement of free triiodothyronine (fT3) in serum to assess thyroid hormone availability.
  Unit of Measure: Picomoles per liter (pmol/L)
Change in Serum free thyroxine (fT4) levels | At baseline and during follow-up (up to 5 years)
  Measurement of free thyroxine (fT4) in serum to assess thyroid hormone production and metabolic status.
  Unit of Measure: Picomoles per liter (pmol/L)
Change in Timed Up and Go (TUG) test | At baseline and during follow-up (up to 5 years)
  Assessment of functional mobility using the Timed Up and Go (TUG) test. Participants will be instructed to rise from a seated position, walk 3 meters, turn around, walk back to the chair, and sit down. The time taken to complete the test will be measured with a stopwatch. Longer times indicate reduced mobility and higher risk of falls. Unit of Measure:
  Seconds (s)
Change in sperm vitality (Eosin-nigrosin test, male patients) | At baseline and during follow-up (up to 5 years)
  Assessment of sperm vitality using the eosin-nigrosin staining test. Semen samples will be stained and analyzed microscopically to distinguish live (unstained) from dead (stained) spermatozoa. The percentage of live spermatozoa will be recorded.
  Unit of Measure:
  Percentage of live spermatozoa (%)
Serum levels of pro-inflammatory and anti-inflammatory cytokines | At baseline and during follow-up (up to 5 years)
  Quantification of circulating pro-inflammatory cytokines using ELISA, including: interleukin-1 beta (IL-1β); interleukin-6 (IL-6); and tumor necrosis factor-alpha (TNF-α). These biomarkers will be used to assess systemic inflammatory status. Quantification of anti-inflammatory cytokines via ELISA, including: interleukin-10 (IL-10) and interleukin-1 receptor antagonist (IL-1Ra), to evaluate immune-regulatory balance. Measurement of additional inflammatory mediators including: interleukin-8 (IL-8), monocyte chemoattractant protein-1 (MCP-1), and interferon-gamma (IFN-γ) using ELISA-based quantification.
  Unit of Measure: Picograms per milliliter (pg/mL)
Serum levels of adipokines and other adiposity-related biomarkers | At baseline and during follow-up (up to 5 years)
  Quantification of circulating adipokines involved in metabolic regulation using ELISA, including: leptin; adiponectin; and resistin. These biomarkers will be analyzed in relation to body composition and inflammatory status. Measurement of additional adipose tissue-derived biomarkers using ELISA, including: visfatin; chemerin; and omentin. These markers will be evaluated for their association with inflammation, insulin resistance, and metabolic dysfunction.
  Unit of Measure: Nanograms per milliliter (ng/mL)
Gene expression of markers of HPA axis activity and glucocorticoid sensitivity | At baseline and during follow-up (up to 5 years)
  Quantification of mRNA expression levels of selected genes involved in hypothalamic-pituitary-adrenal (HPA) axis regulation and glucocorticoid responsiveness. Target genes include, but are not limited to: FKBP5, FKBP4, NR3C1 (glucocorticoid receptor), CRH, CRHR1, POMC, and PER1. Gene expression will be assessed in peripheral blood mononuclear cells (PBMCs) using RT-qPCR/NanoString-based methods. Relative expression levels will be normalized to reference genes and analyzed for treatment-related variation.
  Unit of Measure:
  Relative expression level (fold change from baseline)

OTHER OUTCOMES:
Availability of biological samples for future biomarker analyses | Samples collected at baseline and follow-up; stored until the end of the study (5 years)
  Description: Plasma, serum, and urine samples will be biobanked for future exploratory analyses, including gene expression, cytokines, miRNAs, hormones, and other circulating factors. These analyses will be exploratory.
  Unit of Measure: Not applicable (biological samples only)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Experimental Medicine, Sapienza University of Rome, Rome, Italy, Italy

REFERENCES:
- [Background] Sytkowski PA, Kannel WB, D'Agostino RB. Changes in risk factors and the decline in mortality from cardiovascular disease. The Framingham Heart Study. N Engl J Med. 1990 Jun 7;322(23):1635-41. doi: 10.1056/NEJM199006073222304. PMID 2288563
- [Background] Cantisani V, Bertolotto M, Weskott HP, Romanini L, Grazhdani H, Passamonti M, Drudi FM, Malpassini F, Isidori A, Meloni FM, Calliada F, D'Ambrosio F. Growing indications for CEUS: The kidney, testis, lymph nodes, thyroid, prostate, and small bowel. Eur J Radiol. 2015 Sep;84(9):1675-84. doi: 10.1016/j.ejrad.2015.05.008. Epub 2015 May 14. PMID 26014102
- [Background] Pozza C, Gianfrilli D, Fattorini G, Giannetta E, Barbagallo F, Nicolai E, Cristini C, Di Pierro GB, Franco G, Lenzi A, Sidhu PS, Cantisani V, Isidori AM. Diagnostic value of qualitative and strain ratio elastography in the differential diagnosis of non-palpable testicular lesions. Andrology. 2016 Nov;4(6):1193-1203. doi: 10.1111/andr.12260. Epub 2016 Aug 27. PMID 27565451
- [Background] Auchus RJ, Hamidi O, Pivonello R, Bancos I, Russo G, Witchel SF, Isidori AM, Rodien P, Srirangalingam U, Kiefer FW, Falhammar H, Merke DP, Reisch N, Sarafoglou K, Cutler GB Jr, Sturgeon J, Roberts E, Lin VH, Chan JL, Farber RH; CAHtalyst Adult Trial Investigators. Phase 3 Trial of Crinecerfont in Adult Congenital Adrenal Hyperplasia. N Engl J Med. 2024 Aug 8;391(6):504-514. doi: 10.1056/NEJMoa2404656. Epub 2024 Jun 1. PMID 38828955
- [Background] Whitaker MJ, Huatan H, Ross RJ. Chronotherapy based on modified-release hydrocortisone to restore the physiological cortisol diurnal rhythm. Drug Deliv Transl Res. 2023 Jan;13(1):1-8. doi: 10.1007/s13346-022-01183-w. Epub 2022 May 26. PMID 35618893
- [Background] Schroder MAM, Claahsen-van der Grinten HL. Novel treatments for congenital adrenal hyperplasia. Rev Endocr Metab Disord. 2022 Jun;23(3):631-645. doi: 10.1007/s11154-022-09717-w. Epub 2022 Feb 23. PMID 35199280
- [Background] Merke DP, Mallappa A, Arlt W, Brac de la Perriere A, Linden Hirschberg A, Juul A, Newell-Price J, Perry CG, Prete A, Rees DA, Reisch N, Stikkelbroeck N, Touraine P, Maltby K, Treasure FP, Porter J, Ross RJ. Modified-Release Hydrocortisone in Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2063-e2077. doi: 10.1210/clinem/dgab051. PMID 33527139
- [Background] Pivonello R, Isidori AM, De Martino MC, Newell-Price J, Biller BM, Colao A. Complications of Cushing's syndrome: state of the art. Lancet Diabetes Endocrinol. 2016 Jul;4(7):611-29. doi: 10.1016/S2213-8587(16)00086-3. Epub 2016 May 10. PMID 27177728
- [Background] Stikkelbroeck NM, Otten BJ, Pasic A, Jager GJ, Sweep CG, Noordam K, Hermus AR. High prevalence of testicular adrenal rest tumors, impaired spermatogenesis, and Leydig cell failure in adolescent and adult males with congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2001 Dec;86(12):5721-8. doi: 10.1210/jcem.86.12.8090. PMID 11739428
- [Background] Falhammar H, Nystrom HF, Ekstrom U, Granberg S, Wedell A, Thoren M. Fertility, sexuality and testicular adrenal rest tumors in adult males with congenital adrenal hyperplasia. Eur J Endocrinol. 2012 Mar;166(3):441-9. doi: 10.1530/EJE-11-0828. Epub 2011 Dec 9. PMID 22157069
- [Background] Isidori AM, Venneri MA, Graziadio C, Simeoli C, Fiore D, Hasenmajer V, Sbardella E, Gianfrilli D, Pozza C, Pasqualetti P, Morrone S, Santoni A, Naro F, Colao A, Pivonello R, Lenzi A. Effect of once-daily, modified-release hydrocortisone versus standard glucocorticoid therapy on metabolism and innate immunity in patients with adrenal insufficiency (DREAM): a single-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Mar;6(3):173-185. doi: 10.1016/S2213-8587(17)30398-4. Epub 2017 Dec 8. PMID 29229498
- [Background] Danilowicz K, Bruno OD, Manavela M, Gomez RM, Barkan A. Correction of cortisol overreplacement ameliorates morbidities in patients with hypopituitarism: a pilot study. Pituitary. 2008;11(3):279-85. doi: 10.1007/s11102-008-0126-2. PMID 18459045
- [Background] Schulz J, Frey KR, Cooper MS, Zopf K, Ventz M, Diederich S, Quinkler M. Reduction in daily hydrocortisone dose improves bone health in primary adrenal insufficiency. Eur J Endocrinol. 2016 Apr;174(4):531-8. doi: 10.1530/EJE-15-1096. Epub 2016 Jan 25. PMID 26811406
- [Background] Filipsson H, Monson JP, Koltowska-Haggstrom M, Mattsson A, Johannsson G. The impact of glucocorticoid replacement regimens on metabolic outcome and comorbidity in hypopituitary patients. J Clin Endocrinol Metab. 2006 Oct;91(10):3954-61. doi: 10.1210/jc.2006-0524. Epub 2006 Aug 8. PMID 16895963
- [Background] Pofi R, Ji X, Krone NP, Tomlinson JW. Long-term health consequences of congenital adrenal hyperplasia. Clin Endocrinol (Oxf). 2024 Oct;101(4):318-331. doi: 10.1111/cen.14967. Epub 2023 Sep 7. PMID 37680029
- [Background] Bornstein SR, Allolio B, Arlt W, Barthel A, Don-Wauchope A, Hammer GD, Husebye ES, Merke DP, Murad MH, Stratakis CA, Torpy DJ. Diagnosis and Treatment of Primary Adrenal Insufficiency: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 Feb;101(2):364-89. doi: 10.1210/jc.2015-1710. Epub 2016 Jan 13. PMID 26760044
- [Background] El-Maouche D, Arlt W, Merke DP. Congenital adrenal hyperplasia. Lancet. 2017 Nov 11;390(10108):2194-2210. doi: 10.1016/S0140-6736(17)31431-9. Epub 2017 May 30. PMID 28576284